CLINICAL TRIAL: NCT06108024
Title: Randomized Double-Blind Vehicle-Controlled Study of the Safety and Efficacy of SM-020 Gel 1.0% in Subjects With Seborrheic Keratosis
Brief Title: A Trial to Evaluate the Safety and Efficacy of SM-020 Gel 1.0% in Subjects With Seborrheic Keratosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-213
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SM-020 gel 1.0% (Active Comparator): SM-020 gel 1.0% will be applied topically. Subjects will be treated with twice daily application to 5 to 10 SKTLs for approximately 28 days.
  Interventions: Drug: SM-020 gel 1.0%
- Vehicle gel (Placebo Comparator): Vehicle gel will be applied topically. Subjects will be treated with twice daily application to 5 to 10 SKTLs for approximately 28 days.
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: SM-020 gel 1.0% — SM-020 gel 1.0% will be applied topically. Subjects will be treated with twice daily application to 5 to 10 SKTLs for approximately 28 days.
  Arms: SM-020 gel 1.0%
Drug: Vehicle gel — Vehicle gel will be applied topically. Subjects will be treated with twice daily application to 5 to 10 SKTLs for approximately 28 days.
  Arms: Vehicle gel

SUMMARY:
The objective of the trial is to evaluate the safety and efficacy of SM-020 gel 1.0% in subjects with Seborrheic Keratosis (SK) compared to vehicle gel. It is a randomized, double-blind, vehicle-controlled trial. Approximately 60 subjects will be enrolled. Subjects will apply their assigned investigational product twice daily for 4 consecutive weeks. Subjects will be followed for 12-weeks post final application for a total of approximately 16-weeks of required participation in the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. Must be able to comprehend and willing to sign an informed consent form (ICF).
2. Must complete a signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of the subject's individually identifiable health information.
3. Must be at least 18 years of age.
4. Must have a minimum of 5 eligible facial, truncal, intertriginous, or extremity SKTLs. A maximum of 10 SKTLs will be targeted for treatment. An eligible SKTL must :

   1. Have one or more of the following clinical features throughout the entirety of the lesion consistent with SKs: stuck-on, sharply demarcated, warty, waxy, scaly, milia-like cyst, tan to black
   2. For subjects randomized for eligibility assessment with dermoscopy, SKs must also have one or more of the following dermoscopy features throughout the entirety of the lesion: crypts (comedo-like openings), milia cysts, hairpin vessels with white halo, sharp demarcation, blue-white pigmentation/veil as long as milia and crypts are present within, more than one color, cerebriform structure (network-like pattern/gyri and sulci/ridges and fissures/fat fingers), irregular vessels (inframammary only), granularity at periphery, stalactite/Tsingy pattern, plate-like/fractured pattern (Simionescu et al., 2012)
   3. Have a Physician's Lesion Assessment (PLA) of 2 (a thickness that is ≤1mm)
   4. Have a greatest diameter that is >5mm but ≤15mm
   5. Be a discrete, well-defined, separate lesion
   6. Not be covered with hair which, in the Investigator's opinion, would interfere with the study gel treatment or the study evaluations
   7. Not be pedunculated
   8. Not be on the eyelid
   9. Not be within 5mm of the orbital rim
5. Must be free of any known disease state or physical condition which, in the Investigator's opinion, might impair evaluation of any SKTL or which exposes the subject to an unacceptable risk by study participation.
6. Must be willing and able to follow all study instructions and to attend all study visits.
7. Must be willing to have all partial, incompletely, or non-responding SKTLs removed surgically by shave excision during the final visit.

Exclusion Criteria:

Subjects meeting any of the following criterion will be ineligible and excluded from this study:

1. Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control (such as oral contraceptive pills (OCPs), Intrauterine devices (IUDs), birth control implants, vaginal rings, or injections) for the duration of the study.
2. SK lesions that are clinically atypical and/or rapidly growing in size or number.
3. SK lesions that have any of the following features indicative of malignancy under dermoscopy: pinpoint vessels, smooth blue-white pigmentation/veil without milia or crypts within, hairpin vessels without white halo, white artifacts, irregular vessels (except for inframammary lesions). Additionally, for lesions randomized to dermoscopy, SK lesions must not have a moth-eaten border or fingerprint structures indicative of lentigos or a network pattern indicative of a melanocytic lesion.
4. Presence of multiple eruptive SK lesions (sign of Leser-Trelat).
5. Current systemic malignancy.
6. Any use of the following systemic therapies within the specified period, or unwilling to meet the following washouts, prior to the Baseline visit and while on study:

   1. Retinoids; 180 days
   2. Chemotherapy; 180 days
   3. Immunosuppressive therapy; 28 days
   4. Biologics (e.g., interferon, interferon inducers, or immunomodulators); 28 days
   5. Glucocorticosteroids; 28 days
   6. Anti-metabolites (e.g., methotrexate); 28 days
   7. Vismodegib; 180 days
   8. Known photosensitizing medications or CYP3A inducers/inhibitors; 28 days
7. Any use of the following topical therapies within the specified period, or unwilling to meet the following washouts, prior to the Baseline visit and while on study, on or in a proximity to any SKTL that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   1. Laser, light or other energy-based therapy [e.g., intense pulsed light (IPL), photo-dynamic therapy (PDT)]; 180 days
   2. Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-fluorouracil, or ingenol mebutate; 60 days
   3. Retinoids; 28 days
   4. Microdermabrasion or superficial chemical peels; 14 days
   5. Glucocorticosteroids or antibiotics; 14 days
8. Occurrence or presence of any of the following within the specified period prior to the Baseline visit on or in the proximity of any SKTL that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   1. Cutaneous malignancy; 180 days
   2. Sunburn; currently
   3. A pre-malignancy (e.g., actinic keratosis); currently
   4. Body art (e.g., tattoos, piercing, etc.); currently
9. History of sensitivity to any of the ingredients in the investigational product.
10. Any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or other condition(s) (e.g., sunburn, excessive hair, open wounds, lupus, photosensitive disorders etc.) that, in the opinion of the Investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
11. Participation in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to the Screening visit.
12. History of hypertrophic scarring or keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Superiority of active over vehicle as measured by the proportion of all SKTLs (Seborrheic Keratosis Target Lesion) that achieve a PLA score of 0 | Screening, Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, and Week 16
  The PLA is an Investigator assessment of SK lesion severity based on presence of SK and the thickness of the SK lesion. The PLA will be determined for each SKTL at all clinic study visits from Visit 1/Screening to Visit 9/Last Visit.
  Physician's Lesion Assessment Grade Descriptor
  0 Clear: no visible seborrheic keratosis lesion
  1. Near Clear: a visible seborrheic keratosis lesion with a surface appearance different from the surrounding skin (not elevated)
  2. Thin: a visible seborrheic keratosis lesion (thickness ≤1mm)
  3. Thick: a visible seborrheic keratosis lesion (thickness >1mm)
Safety and Tolerability as evaluated by assessment of the severity of the signs and symptoms of Application Site Reactions (ASRs) of Seborrheic Keratosis | Through week 16 (Visit 9)
  Application site reactions will be evaluated based on the scores for erythema, edema, exudation, erosion/ulceration, hyperpigmentation, and hypopigmentation by the Investigator, and the additional symptoms of pain, burning, stinging, and pruritus. Scale 0=None, 1=slight, 2=Moderate, 3=Significant with 0 being the minimum value and 3 being the maximum value, with a higher value indicating higher severity.
Safety and Tolerability as evaluated by review of adverse events | Through week 16 (Visit 9)
  Grade 1 = Mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL Grade 3 = Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL Grade 4 = Life-threatening consequences: urgent intervention indicated Grade 5 = Death related to AE with Grade 1 being the minimum value and Grade 5 being the maximum value, with a higher value indicating higher severity.

SECONDARY OUTCOMES:
Superiority of active over vehicle as measured by the percentage of facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs that achieve clearance (PLA score of 0) | Through week 16
  The Physician's Lesion Assessment (PLA) is an Investigator assessment of SK lesion severity based on presence of SK and the thickness of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.
Superiority of active over vehicle as measured by the percentage of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs with a PLA of 0 or 1 | Through week 16
  The Physician's Lesion Assessment (PLA) is an Investigator assessment of SK lesion severity based on presence of SK and the thickness of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.
Superiority of active over vehicle, based on the time to all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs achieving a PLA of 0 | Through week 16
  The Physician's Lesion Assessment (PLA) is an Investigator assessment of SK lesion severity based on presence of SK and the thickness of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.
Superiority of active over vehicle as measured by the percentage of subjects achieving clearance of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs | Through week 16
Superiority of active over vehicle as measured by the percentage of subjects achieving clearance of at least 60% of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLS, and extremity SKTLs | Through week 16
Superiority of active over vehicle as measured by the percentage of all SKTLs/subject, facial SKTLs/subject, truncal SKTLs/subject, intertriginous SKTLs/subject, and extremity SKTLs/subject achieving a PLA of 0 | Through week 16
  The Physician's Lesion Assessment (PLA) is an Investigator assessment of SK lesion severity based on presence of SK and the thickness of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.
Superiority of active over vehicle as measured by the percentage of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs with a SSA (Subject's Self-Assessment) of 0 or 1 | Through week 16
  The SSA is a subject's self-reported assessment of SK lesion severity based on presence of SK and the thickness and coloration of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.
Superiority of active over vehicle as measured by the percentage of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs with a SSA of 0 | Through week 16
  The SSA is a subject's self-reported assessment of SK lesion severity based on presence of SK and the thickness and coloration of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.
Superiority of active over vehicle as measured by the percent recurrence of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs | Through week 16
  The SSA is a subject's self-reported assessment of SK lesion severity based on presence of SK and the thickness and coloration of the SK lesion. The minimum value is 0 and the maximum value is 3 with a higher value indicating higher severity or significance.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Driven Research LLC, Coral Gables, Florida
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon